CLINICAL TRIAL: NCT04049396
Title: The Effect of Berberine on Lipid Profile, Liver Enzymes and Fasting Blood Glucose in Patients With Non-Alcoholic Fatty Liver Disease (NAFLD): A Randomized Controlled Trial
Brief Title: Berberine and Non-Alcoholic Fatty Liver Disease (NAFLD)
Acronym: NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lida Nejati (Other)
Responsible Party: Sponsor-Investigator, Lida Nejati, Senior Nutritionist, MSc of Nutrition, Science and Research Branch, Islamic Azad University, Tehran, Iran, Islamic Azad University, Sanandaj
Organization: Islamic Azad University, Sanandaj (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR.IAU.SRB.REC
Record Dates: First submitted 2019-07-21; First posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD, Berberine, ALP, AST, ALT, FBS, HDL,LDL
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Berberine

STUDY DESIGN:
Intervention Model Description: In this study , samples were randomly divided into two groups receiving and not receiving supplement
Masking Description: This study was conducted as an open-label, randomized controlled trial .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berberine (Experimental): Berberine (6.25 g/day)
  Interventions: Other: Berberine
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Berberine — 24 Patient consumed 6,25 g/day Berberine for 6 weeks
  Arms: Berberine

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD), one of the most common liver dysfunctions, affects about one-fourth of the global adult population and has a significant mortality rate between 6.3% and 33%.NAFLD can lead to other serious illnesses. The disease is associated with a group of metabolic comorbid conditions, including type 2 diabetes mellitus (T2DM), obesity, hypertension, and hyper-cholesterolemia, which are potential risk factors for progressive liver disease.This study sought to evaluate the therapeutic effect of berberine on the liver function and metabolic profiles of patients with NAFLD. In this context,A six week, open-label randomized controlled trial was conducted in a single medical center at Takestan Hospital, Iran. A total of 281 patients with NAFLD were enrolled and randomly assigned to treatment arm with (n=24) or without (n=24) berberine. All patients had received pre-randomization lifestyle training including recommendations on low-fat diet. Blood examinations were performed to evaluate glucose, lipid profile, and liver enzymes both at the beginning of the study and upon the completion of the trial (day 45). To assess tolerability of the study intervention and any possible adverse events, patients in both groups were required to attend weekly follow-up visits.

DETAILED DESCRIPTION:
A seven-week (45-day), open-label, randomized controlled trial was conducted in a medical center affiliated with the Ministry of Welfare and Social Security in Iran to study the impact of berberine on liver function and metabolic profiles of patients with NAFLD. Hospital employees who met the enrollment criteria were identified through electronic health records (EHRs) available in a human resource database of employee routine annual examinations. Using a computer-generated random-allocation sequence, eligible employees were equally assigned (1:1) to berberine 6.25 g per day (arm A) or no intervention (Arm B). Berberine was administered orally (100 g dried berberine in 5 Liter water boiled at 167°F until 4Liter).). To control the potential impact of confounders on outcome measures, and to balance the daily dietary and physical activity among the study groups, all participants were trained by skilled experts on lifestyle and behavior improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an age range between 18 to 65 years(inclusive).
* Patients with Liver fat content assessed by MRS≥13%.
* Patients must meet the criteria for impaired glucose regulation
* Course of diabetic mellitus less than 1 year
* Informed consent signed

Exclusion Criteria:

* Any causes of chronic liver disease other than NAFLD(such as-but not restricted to- alcohol or drug abuse, medication, chronic hepatitis B or C, autoimmune, etc.);

  * Patients with significantly impaired liver function: ALT or AST≥2 times upper limit of normal;
  * Patients with type 1 diabetes mellitus or gestational diabetes or special type diabetes;
  * Course of diabetes more than 1 years;
  * Diabetics patients who have taken or are taking oral glucose-lowering drugs or insulin;
  * Diabetics patients with a HbA1c>7.5% on initial visit;
  * Patients with severe diabetes complications(diabetes ketoacidosis, diabetes coma or with symptomatic of diabetes coma; dysfunction of nerve, retinopathy, dysfunction of kidney);
  * Patients with a history of clinically significant heart disease(myocardial infarct, heart failure, and/or severe cardiac rhythm);
  * Complicating severe infection,within 6 months after operation, severe trauma;
  * Patients with excess alcohol consumption≥140g/week(male); ≥70g/week(female);
  * Patients have participated other clinical trials within 24 weeks;
  * Patients with a history of drug allergy to berberine;
  * Patients with gestation or possible gestation or lactation, or males or females expecting gestation during clinical trial;
  * Mental diseases patients;
  * Those who refuse to sign informed consent;
  * Any other conditions, which, in the opinion of the investigators would impede competence or compliance or possibility of hindering completion of the study;
  * Patients with serum triglyceride≥5.0mmol/L;
  * Patients with thyroid disease, including hyperthyroidism or hypothyroidism.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Alanine Aminotransferase (ALT) | Baseline and 6 weeks after
  Serum Alanine Aminotransferase concentration (units per liter)
Change from baseline of Aspartate Aminotransferase (AST) | Baseline and 6 weeks after
  Serum Aspartate Aminotransferase concentration(units per liter)
Change from baseline of Alkaline Phosphatase( ALP) | Baseline and 6 weeks after
  Serum Alkaline Phosphatase concentration (units per liter)

SECONDARY OUTCOMES:
Change from baseline of fasting blood sugar(FBS) | Baseline and 6 weeks after
  Fasting blood sugar concentration (mg/dl)
Change from baseline of total cholesterol (TC) | Baseline and 6 weeks after
  Serum total cholesterol concentration (mg/dl)
Change from baseline of LDL-Cholesterol | Baseline and 6 weeks after
  Serum LDL-Cholesterol concentration (mg/dl)
Change from baseline of HDL - Cholesterol | Baseline and 6 weeks after
  Serum HDL-Cholesterol concentration (mg/dl)
Change from baseline of Triglyceride (TG) | Baseline and 6 weeks after
  Serum Triglyceride concentration (mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Sciences & Research Branch,Azad University of Tehran, Tehran, Iran